CLINICAL TRIAL: NCT01151579
Title: Prospective Trial of Effect of Nebulized Bronchodilators on Heart Rate and Arrhythmias in Critically Ill Adult Patients
Brief Title: Effect of Nebulized Bronchodilators on Heart Rate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fahim Khorfan, MD (Industry)
Collaborators: Ascension Health (Industry)
Responsible Party: Sponsor-Investigator, Fahim Khorfan, MD, ICU Pulmonologist, Ascension Health
Organization: Ascension Health (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: ME 07-0011
Record Dates: First submitted 2010-06-24; First posted 2010-06-28 (Estimated); Results first posted 2015-10-23 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-09

CONDITIONS: COPD; Sepsis; Shock
Keywords: Tachycardia; tachyarrhythmias; bronchodilator therapy; Critically ill patients
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Sepsis; Shock; Tachycardia | interventions — Levalbuterol; Ipratropium; Albuterol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levalbuterol 0.63 (Active Comparator): Patients received an initial dose of levalbuterol 0.63 mg alternating with albuterol 2.5 mg.
  Interventions: Drug: Levalbuterol; Drug: Albuterol
- Levalbuterol 1.25 (Active Comparator): Patients received an initial dose of levalbuterol 1.25 mg alternating with albuterol 2.5 mg.
  Interventions: Drug: Levalbuterol; Drug: Albuterol

INTERVENTIONS:
Drug: Levalbuterol — inhaled Levalbuterol 0.625 mg inhaled Levalbuterol 2.5 mg
  Other Names: Xopenex; ipratropium
Drug: Albuterol — Nebulized albuterol 2.5mg
  Other Names: Salbutamol

SUMMARY:
The purpose of the study is to determine adverse events rates of nebulized albuterol versus levalbuterol among adult critically ill patients and determine if a differential exists in adverse events between the two drugs.

DETAILED DESCRIPTION:
A randomized, single-blind, cross-over, prospective study was conducted in seventy critically ill adult patients with acute air flow obstruction. Patients were randomized to nebulized albuterol alternating with levalbuterol every 4 to 6 hours. Group A received albuterol 2.5 mg alternating with levalbuterol 0.63 mg. Group B received albuterol 2.5 mg alternating with levalbuterol 1.25 mg. All patients received nebulized ipratropium bromide 500 micrograms with each treatment. Heart rate and cardiac rhythm were continuously recorded before and 15 minutes after finishing each treatment. Any new rhythm abnormalities between treatments were also recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adults who required inhaled bronchodilator therapy in the form of short acting beta adrenergic receptor agonist and short acting anti-cholinergic treatment every 4-6 hours for respiratory functions

Exclusion Criteria:

* Known allergy or sensitivity to study medications
* Baseline heart rate was greater than 110 beats per minute

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2008-12; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fahim Khorfan, MD, Principal Investigator — Ascension Health; Kimberly R Barber, PhD, Study Director — Ascension Health
Locations (1):
- Genesys Regional Medical Center, Grand Blanc, Michigan, United States

REFERENCES:
- [Derived] Khorfan FM, Smith P, Watt S, Barber KR. Effects of nebulized bronchodilator therapy on heart rate and arrhythmias in critically ill adult patients. Chest. 2011 Dec;140(6):1466-1472. doi: 10.1378/chest.11-0525. Epub 2011 Sep 29. PMID 21960699

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began initially August 21, 2007 at the medical center ICU.
Pre-assignment Details: Patients were excluded if they had a known allergy or sensitivity to study medications or if baseline heart rate was greater than 110 bpm. Treating physicians detremined the need for and frequency of treatment with bronchodilator therapy. All other medications were allowed.
Groups:
- Nebulized Albuterol 2.5mg: Patients were randomized to receive an initial dose of albuterol 2.5 mg alternating with levalbuterol 0.63 mg.
Period: Overall Study
Arm/Group | Nebulized Albuterol 2.5mg | Levalbuterol 1.25
Started | 58 | 31
Completed | 46 | 24
Not Completed | 12 | 7
Not completed — Physician Decision | 3 | 1
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Not meet inclusion criteria | 6 | 4

BASELINE CHARACTERISTICS:
Population: The number analyzed was determined by the power calculation and based on the number of participants randomized to treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nebulized Albuterol 2.5mg | Levalbuterol 1.25 | Total
Number analyzed (Participants) | 58 | 31 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 9 | 27
  >=65 years | 40 | 22 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (13.1) | 67.5 (13.7) | 67.3 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 12 | 43
  Male | 27 | 19 | 46
Region of Enrollment [Number; unit: participants]
  United States | 58 | 31 | 89

OUTCOME MEASURES:

1. Primary Outcome: Heart Rate in Beats Per Minute
Description: Average difference in Heart rate between pre and post breathing treatments
Time Frame: Five days
Population: Average change in heart rate from baseline to final breathing treatment.
Measure: Mean (Standard Deviation); unit: bpm
Units Other Than Participants: Breathing treatment episodes
Arm/Group | Nebulized Albuterol 2.5mg | Levalbuterol 1.25
Number analyzed (Participants) | 46 | 24
Number analyzed (Breathing treatment episodes) | 604 | 232
bpm | -0.16 (5.1) | 1.40 (5.4)
Statistical Analysis 1: Comparison: Nebulized Albuterol 2.5mg vs Levalbuterol 1.25; Null Hypothesis: No difference between groups in heart rate changes from baseline following treatment. Sample size calculation determined a need for at least 400 breathing treatments among 65 patients; Test type: Non-Inferiority or Equivalence — A total of at least 400 treatemnts or 65 patients was required to achieve 94% power to determine a 1% change by treatment or a 5% change between groups to be significant at p-value of 0.01 and o.05, respectively; p = 0.01, Mixed Models Analysis; Mean Difference (Final Values) = 1, Standard Error of Mean 0.5

2. Secondary Outcome: Arrhythmias
Description: Any new arrhythmia documented in the medical record that occurred between breathing treatments.
Time Frame: 15 minutes after each treatment for average of 3 to 5 days
Population: The percentage of arrhythmias among the number of breathing treatments.
Measure: Number; unit: percent
Arm/Group | Nebulized Albuterol 2.5mg | Levalbuterol 1.25
Number analyzed (Participants) | 46 | 24
percent | 0.33 | 1.3
Statistical Analysis 1: Comparison: Nebulized Albuterol 2.5mg vs Levalbuterol 1.25; Null hypothesis: no difference in incidence of arrhythmias between groups within the total number of breathing treatments; Test type: Superiority or Other; p = 0.05, Chi-squared — Analysis adjusted with Fischer exact chi-square for rare occurrences; Risk Ratio (RR) = 1

3. Secondary Outcome: Total Number of Participants With Arrhythmias
Description: Documented new arrhythmia occurring during study.
Time Frame: Five days
Population: Number of patients for whom arrhythmias occurred within 5 days after treatment initiation.
Measure: Number; unit: participants
Arm/Group | Nebulized Albuterol 2.5mg | Levalbuterol 1.25
Number analyzed (Participants) | 46 | 24
participants | 2 | 3
Statistical Analysis 1: Comparison: Nebulized Albuterol 2.5mg vs Levalbuterol 1.25; To report on the number of events; Test type: Superiority or Other; p = 0, descriptive; Descriptive statistics (frequency) used to report the number of participants experiencing an event

ADVERSE EVENTS:
Time Frame: Within 5 days of treatment initiation and within 15 minutes of each individual treatment.
Description: Cardiac arrhythmia
Arm/Group | Nebulized Albuterol 2.5mg | Levalbuterol 1.25
Serious Adverse Events (participants affected / at risk) | 2/58 | 3/31
Other Adverse Events (participants affected / at risk) | 0/58 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nebulized Albuterol 2.5mg (N=58) | Levalbuterol 1.25 (N=31)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 3 (3) — Cardiac arrhythmia as documented by healthcare provider.

LIMITATIONS AND CAVEATS:
Potential limitations are its single-center site and that the design may not have adequately eliminated all carryover effects from the levalbuterol. However, the number of side effects without carryover would be even lower than we observed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes